CLINICAL TRIAL: NCT03619668
Title: Chemo-radiotherapy as Main Treatment Strategy for Rectal Cancer. Can we Provide a More Precise and Effective Treatment
Acronym: AMPERE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Dennis Tideman Arp, Medical Physicist, Aalborg University Hospital
Other Study IDs: N-20170064
Record Dates: First submitted 2018-06-29; First posted 2018-08-08 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Rectal Cancer; Rectal Adenocarcinoma; Locally Advanced Malignant Neoplasm
Keywords: Effect of radiotherapy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this project is to obtain important information about the tumour and surrounding organs during preoperative chemo-radiotherapy for patients with adenocarcinoma of the rectum. The knowledge generated in this project has the potential to make future radiotherapy treatments (RT) of rectal cancer patients more precise, with less side effects. This could lead the way to make chemo-radiotherapy the main treatment modality and spare a large group of patients from the risk of severe complications after surgery. Specifically, we aim to obtain:

* A characterization of systematic and random changes in position and shape of tumours and surrounding organs during RT.
* A patient-specific pre-treatment characterization of random uncertainties in position and shape of the tumour during radiotherapy. This will be used to create and assess an individual, patient-specific treatment strategy, with the possibility to implement an adaptive RT strategy using the information obtained from the MRI-scans during treatment.
* Information about treatment response and local toxicity from morphological and functional data before, during and after CRT.

DETAILED DESCRIPTION:
Patients diagnosed with locally advanced adenocarcinoma of the rectum are treated with concomitant chemo-radiotherapy (CRT), with the aim of reducing local recurrences. Depending on tumor location, this is a pre-operative procedure prior to total mesorectal excision or partial mesorectal excision. The surgery is associated with a high risk of postoperative morbidity, however, especially when combined with CRT. Consequently, recent years have seen an increasing focus on other therapeutic approaches, such as "watch and wait", where the aim is to treat some patients with definitive CRT alone. The success of these new approaches directly relies on the effectiveness of the radiotherapy (RT) treatment and thereby on the level as well as the accuracy of the delivered dose to the tumor.

Standard treatment today is based on a single set of CT- and MRI-scans, which are insufficient to estimate the organ motion during RT. Precise knowledge about the variation in position and shape of the tumor using multiple MRI scans before and during RT will have the potential to make future radiotherapy treatments more precise with less side effects.

The investigators will conduct a prospective study of sequential MRI scans before and during CRT. Patients will be MRI scanned six times in addition to the standard MRI-scan appointments and follow-up. This will provide a total of 9 MRI-scans of each patient; 3 before RT, 3 during RT and 3 during follow up. The information gained from these additional scans will provide a much better understanding of the tumor and organs during RT.

This project's overall focus is to make future RT treatments of rectal cancer patients as precise and efficient as possible. This could contribute to and aid the paradigm shift of making chemo-radiotherapy the main treatment strategy for some rectal cancer patients. This has the potential to spare patients of the severe morbidities associated with surgery, as well as the need for stomas.

ELIGIBILITY:
Inclusion Criteria:

All patients referred to standard chemoradiotherapy for locally advanced rectal cancer.

Exclusion Criteria:

* Prior surgery in pelvic minor region
* Pacemaker
* Neurostimulator
* Other non MR-compatible implants
* Pregnancy
* Incapable of undergoing MRI
* Incapable of understanding the patient information
* Allergic to contrast agent
* Contraindication for Buscopan
* Reduced renal function (GFR < 50 ml/min) Patients who cannot tolerate the contrast used for DCE-MRI (due to allergies, contraindications for Buscopan or reduced renal function (GFR < 50 ml/min)) will still be offered inclusion in the study, but without the contrast-based MRI scans.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to standard chemoradiotherapy for locally advanced rectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Changes in position and shape of the tumour during RT. | Baseline, 3-4 days, an average of 9 days, an average of 16 days, an average of 22 days, average of 37 days
  Use additional MRI scans before radiotherapy (for random changes) and during radiotherapy (for systematic changes). The gross tumor volume (GTV), clinical target volume (CTV) will be delineated separately on CT and all MRI-scans. Using a rigid bony anatomy-based method, the MRI-scans will be registered to the planning CT scan, to allow a comparison of the position and shape variations of the volumes. The information gained will be used to evaluate the relevance of current population based planning target volume (PTV) margins, and, if relevant, provide updated recommendations for treatment margins.

SECONDARY OUTCOMES:
Changes in position and shape of organs during RT. | Baseline, 3-4 days, an average of 9 days, an average of 16 days, an average of 22 days, average of 37 days
  Use additional MRI scans before radiotherapy (for random changes) and during radiotherapy (for systematic changes). The organs at risk (OAR) will be delineated separately on CT and all MRI-scans. Using a rigid bony anatomy-based method, the MRI-scans will be registered to the planning CT scan, to allow a comparison of the position and shape variations of the volumes.
Patient specific pre-treatment systematic changes in position and shape of CTV during radiotherapy. | Baseline, 3-4 days, an average of 9 days.
  Will be used to create an individual patient specific CTV-PTV margin.
Change in treated volume using adaptive radiotherapy | Baseline, an average of 7 days, an average of 14 days, average of 28 days
  An adaptive CTV-to-PTV margin will be calculated and the impact on the treated volume of PTV and OARs is assessed.
Change in the functional imaging parameter: ADC-value. | Baseline, 3-4 days, an average of 9 days, an average of 16 days, an average of 22 days, average of 37 days, an average of 1 year, an average of 2 years, an average of 3 years
  MRI scans providing morphological and functional data before, during and after CRT will provide information about treatment response and local toxicity. The ADC-value provided from the diffusion weighted imaging (DWI-) MRI scans will be analysed and compared to the morphological data. The change in the ADC value will be analysed and compared to RT dose plans. These will subsequently be compared to treatment-related adverse events as assessed by CTCAE v4.0 and patient reported outcome as assessed by LARS score and EORTC quality of life questionnaires (QLQ-C30 and QLQ-CR29).
Change in functional imaging parameter: Ktrans. | Baseline, 3-4 days, an average of 9 days, an average of 16 days, an average of 22 days, average of 37 days, an average of 1 year, an average of 2 years, an average of 3 years
  MRI scans providing morphological and functional data before, during and after CRT will provide information about treatment response and local toxicity. The Ktrans-value provided from the dynamic contrast enhanced (DCE-) MRI scans will be analysed and compared to the morphological data. The change in the Ktrans-value will be analysed and compared to RT dose plans. These will subsequently be compared to treatment-related adverse events as assessed by CTCAE v4.0 and patient reported outcome as assessed by LARS score and EORTC quality of life questionnaires (QLQ-C30 and QLQ-CR29).

CONTACTS AND LOCATIONS:
Overall Officials: Dennis T. Arp, Medical Physicist, Principal Investigator — Department of Medical Physics, Oncology, Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

DOCUMENTS (1):
  • Study Protocol (2018-05-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT03619668/Prot_000.pdf